CLINICAL TRIAL: NCT05016284
Title: A Double-blind, Superiority, and Randomized Controlled Trial to Evaluate the Efficacy of a Novel Cannabidiol Cream for Treatment of Atopic Dermatitis
Brief Title: Comparison of JW-100 and EUCRISA for the Treatment of Atopic Dermatitis
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Applied Biology, Inc. (Industry)
Collaborators: Jupiter Wellness, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JW-100-RCT-001
Record Dates: First submitted 2021-08-17; First posted 2021-08-23 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-11

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — crisaborole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JW-100 (Experimental): Subjects applying JW-100 cream twice daily at home (experimental group).
  Interventions: Other: JW-100
- EUCRISA (Active Comparator): Subjects applying EUCRISA® (Pfizer) product twice daily at home (comparator group).
  Interventions: Drug: Eucrisa

INTERVENTIONS:
Other: JW-100 — Cosmetic CBD cream (JW-100)
  Arms: JW-100
Drug: Eucrisa — Topical EUCRISA®, Pfizer
  Arms: EUCRISA

SUMMARY:
To compare the efficacy of a JW-100 cream with active control (commercially available as EUCRISA®, Pfizer) for the treatment of atopic dermatitis (AD) in adult patients with mild to moderate AD measured with the Investigator's Static Global Assessment (ISGA) scale.

DETAILED DESCRIPTION:
Atopic dermatitis (AD) is one of the most common inflammatory skin diseases, affecting 13% of children and approximately 7% of adults in the United States. AD is often stimulated by a cascade of inflammatory events; thus, corticosteroids, immunosuppressive drugs, and antihistamines are often prescribed. Many industrialized countries have legalized botanical cannabis and its extracts for medical purposes. The most clinically relevant components of botanical cannabis are the cannabinoid agents delta-9-tetrahydrocannabinol (THC), cannabidiol (CBD), and the noncannabinoids compounds, terpenoids, and flavonoids. The aim of this study is to explore the efficacy of a novel cannabidiol cream in the treatment of atopic dermatitis in comparison with a commercially available product from Pfizer (EUCRISA®).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years of age.
2. Subject has a clinical diagnosis of stable AD characterized by at least three of the following four features:

   1. Pruritus
   2. Typical morphology and distribution (e.g., flexural lichenification or linearity in adults)
   3. Chronic or chronically-relapsing eczematous/atopic dermatitis
   4. Personal or family history of atopy (i.e., asthma, allergic rhinitis, AD)
3. Subject has an area of AD (excluding the scalp) covering ≥5% and ≤20% body surface area
4. Subject has an Investigator's Static Global Assessment score of 2 or 3
5. If the subject is a woman of childbearing potential, she has a negative urine pregnancy test and agrees to use a protocol approved method of birth control for the duration of the study
6. Subject is non-pregnant and non-lactating
7. Subject is in good general health and free of any known disease state or physical condition which, in the investigator's opinion, might impair evaluation of AD or which exposes the subject to an unacceptable risk by study participation
8. Subject is willing and able to follow all study instructions and to attend all study visits
9. Subject is able to comprehend and willing to sign an Informed Consent Form (ICF)

Exclusion Criteria:

1. Subject has, in the investigator's opinion, spontaneously improving or rapidly deteriorating AD
2. Subject has, in the investigator's opinion, clinically infected AD
3. Subject has any signs or symptoms associated with topical AD therapy (e.g., history of anaphylaxis, hypersensitivity reactions, skin atrophy, striae, pigmentary changes) which, in the investigator's opinion, puts the subject at undue risk by study participation or interfere with the study conduct or evaluations
4. Subject has used any systemic immunosuppressive or immunomodulatory therapy (e.g., etanercept, alefacept, infliximab) with 16 weeks prior to Visit 1
5. Subject has used any phototherapy (e.g., ultraviolet A, ultraviolet B) for AD within four weeks prior to Visit 1
6. Subject has used any systemic AD therapy (e.g., systemic corticosteroids [including intranasal and inhaled corticosteroids at doses >2mg of prednisone or equivalent per day], cyclosporine, immunosuppressants/immunomodulators, Janus Kinase inhibitors, methotrexate, cytostatics) within four weeks prior to Visit 1
7. Subject has used any systemic antibiotics within two weeks prior to Visit 1
8. Subject has used any topical AD therapy (e.g., corticosteroids, calcineurin inhibitors, topical H1 and H2 antihistamines, topical antimicrobials, other medicated topical agents) on the planned treatment area within one week prior to Visit 1
9. Subject is currently using antihistamines (e.g., diphenhydramine, terfenadine) UNLESS the subject has been on a stable dose for at four weeks and agrees to continue that dose for the duration of the study
10. Subject has a history of sensitivity to any of the ingredients in the study medications
11. Subject has any concomitant medical condition which, in the investigator's opinion, might put the subject at undue risk by study participation or interfere with the study conduct or evaluations
12. Subject has participated in an investigational drug trial in which administration of an investigational study medication occurred within 30 days prior to Visit 1.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-11-24 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
The success rate in ISGA score at day 15 with an improvement of grade 2 or greater. | 15 days
  The proportion of patients showing grade 2 or greater improvement using the the Investigator's Static Global Assessment (ISGA) scale.

SECONDARY OUTCOMES:
The success rate of patients with an ISGA score of clear (0) or almost clear (1) at day 15. | 15 days
  The success rate of patients with an ISGA score of clear (0) or almost clear (1) at day 15.
Time to achieve success in ISGA scores 0 and 1. | 15 days
  Time to achieve success in ISGA scores 0 and 1.
Proportion of patients achieving improvement in the severity of the pruritus. | 15 days
  Improvement is defined as reaching scores 0 (none) or 1 (mild), with an improvement greater than or equal to 1 grade from baseline.
Time to improvement in pruritus (scores 0 and 1) | 15 days
  Time to improvement in pruritus (scores 0 and 1)
Percentage mean change from baseline in the severity of AD signs (erythema, exudation, excoriation, induration/papulation, and lichenification). | 15 days
  Percentage mean change from baseline in the severity of AD signs (erythema, exudation, excoriation, induration/papulation, and lichenification).

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Fonseca, MD, Principal Investigator — Hospital Samel
Locations (1):
- Centro Universitário Nilton Lins, Manaus, Amazonas, Brazil

IPD SHARING:
Plan to Share IPD: No
Data will not be shared